CLINICAL TRIAL: NCT00154479
Title: The Correlation Between the Haplotype of Human Leukocyte Antigen (HLA) and Human Papillomavirus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701235
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2006-12-14 (Estimated); Status verified 2003-10

CONDITIONS: Cancer of Cervix
Keywords: Cervical cancer; Human papillomavirus; Human leukocyte antigen; immunologic response; healthy volunteers
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Cervical cancer is the most frequent neoplasm of women in Taiwan and in the world. It influences about 2,700 women with about 1,000 women dying of cervical cancer each year and in Taiwan. Human papillomaviruses (HPV) have been consistently implicated in causing cervical cancer especially those high-risk types which have been strongly associated with cervical cancer. In recent years, there has been compelling evidence that infection with human papillomavirus (HPV) is a major etiologic factor in the development of cervical intraepithelial neoplasia (CIN) and cervical carcinoma.

As in most virus-induced diseases, an adequate immune response is likely to play a key role in the clearance of HPV infections and HPV-related lesions. This assumption is born out by both epidemiological studies and animal models. Immune-compromised patients such as HIV-infected women, organ transplant recipients, and patients suffering from other forms of malignancies, are at a higher risk of developing CIN lesions and invasive cervical cancer. Moreover, several studies establish the existence of natural HPV E7-specific cytotoxic T lymphocyte (CTL) immunity in humans. Only a minority of women infected with oncogenic HPV types develop CIN or cervical cancer. Indeed, the majority of CIN lesions do not progress or even regress to normal cytology, indicating that other factors such as an inadequate immune function are necessary for the development of progressive CIN lesions and cervical carcinoma.

Consequently, the HLA class I and II phenotypes may be correlated with an effective immune response against HPV-associated cervical lesions. Differences in the recognition of foreign antigens, such as those contributed by alleles at the HLA class I or II loci, might be proposed to affect the risk of developing cervical cancer.

In the present proposal, the investigators would like to examine the HLA class I and II associations among Taiwanese women with cervical neoplasia. The purposes of this proposal are:

1. to address the relationships between the HLA class I and II haplotype, HPV infection, and cervical cancer; and
2. to elucidate the immunologic responses to HPV type 16 in different HLA class I and II haplotypes. It will help the investigators to identify which population of HLA genotypes is more susceptible to HPV infection and progresses to invasive cervical cancer. The results of this research will be very useful for the prevention and screening of cervical cancer in the future.

DETAILED DESCRIPTION:
1. To survey the incidence of HPV infection in CIN and cervical cancer patients.

   Using epidemiologic data drawn from a wide range of countries and population groups, investigators have found evidence of HPV in 90% to 95% of cervical cancers. The incidence of HPV in cervical cancer was 79% in our own report. Besides, 91% of high-grade CIN cases and 50% of low-grade CIN cases could be attributed to HPV infection in Taiwanese women. Because these reports for Taiwanese women were published around 10 years ago, it is important to survey and update the incidence of HPV in CIN and cervical cancer patients in Taiwanese women. We will survey the incidence of HPV infection in 500 cervical cancer patients, 100 patients of CIN and 100 normal population patients.
2. To survey the human leukocyte antigen haplotype in CIN and cervical cancer patients.

   HLA class I and II alleles have been reported to associate with the nasopharyngeal carcinoma in Taiwan. Besides, human leukocyte antigen class I and II alleles might interplay in the response to interferon-alpha treatment in Taiwanese patients with chronic hepatitis C virus infection. We will detect the HLA class I and II haplotype first and then correlate them with the CIN and cervical cancer patients.
3. To identify the correlation between HLA class I and II haplotype and HPV infection and CIN and cervical cancer.

   We will further survey the correlation between HLA class I and II and the genotypes of HPV in CIN and cervical cancer patients. We will identify which HLA class I and II haplotypes have positive or negative correlation with HPV infection, CIN and cervical cancer. Then we would determine which specific HLA antigens are important in determining the risk of HPV infection, CIN and cervical cancer.
4. To elucidate the immunologic responses to HPV type 16 in HLA2 with different II haplotypes and the role of immunogenetics in the carcinogenesis of cervical cancer.

HPV type 16 has been identified to be the highest incidence of malignant HPV genotypes in cervical cancer. Our laboratory has set up immunologic assays for evaluating the immune responses to HPV type 16. We will survey the immune response to HPV type 16 in those HLA class I and II haplotypes which have positive or negative correlation with the HPV infection and cervical cancer. We would identify which population of HLA genotype are more susceptible to HPV infection and invasive cervical cancer and elucidate the role of immunogenetics in the HPV infection and carcinogenesis of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Using epidemiologic data drawn from a wide range of countries and population groups, investigators have found evidence of HPV in 90% to 95% of cervical cancers. The incidence of HPV in cervical cancer was 79% in our own report. Besides, 91% of high-grade CIN cases and 50% of low-grade CIN cases could be attributed to HPV infection in Taiwanese women. Because these reports for Taiwanese women were published around 10 years ago. It is important to survey and update the incidence of HPV in CIN and cervical cancer patients in Taiwanese women. We will survey the incidence of HPV infection in 500 cervical cancer patients, 100 patients of CIN and 100 normal population patients.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 2003-10; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Fang Cheng, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Wen-Fang Cheng, Taipei, Taiwan